CLINICAL TRIAL: NCT04929327
Title: Retention Rate of Self-etch Resin Based Sealant With and Without Prior Sandblasting Versus Total Etch Resin Based Sealant in High Caries Risk Patients After One Year Follow up
Brief Title: Retention Rate of Self-etch Resin Based Sealant With and Without Prior Sandblasting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nancy Hussien Abbass Zein El-Abdeen Ebeady, Master's Degree Student- Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CU-5-2021
Record Dates: First submitted 2021-05-30; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Caries; Initial; Pit and Fissure Caries
Keywords: Pit and fissure sealant; Sandblasting; Air abrasion; Retention rate
MeSH Terms: conditions — Van der Woude syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-etch resin based sealant (Active Comparator): Self-etch resin based sealant (prevent seal) without prior sandblasting.
  Interventions: Procedure: Self etch Pit and fissure sealant application (prevent seal)
- Prior Sandblasting (Active Comparator): Self-etch resin based sealant prevent seal) with prior sandblasting.
  Interventions: Procedure: Self etch Pit and fissure sealant application (prevent seal) with prior sandblasting
- Total-etch resin based sealant (Active Comparator): Total-etch resin based sealant (ultraseal XT) (Ultradent Pro. Inc., USA)
  Interventions: Procedure: Total etch resin based sealant ultraseal xt

INTERVENTIONS:
Procedure: Self etch Pit and fissure sealant application (prevent seal) — Sealing deep pits and fissures
  Arms: Self-etch resin based sealant
Procedure: Self etch Pit and fissure sealant application (prevent seal) with prior sandblasting — Sandblasting before Sealing deep pits and fissures
  Arms: Prior Sandblasting
Procedure: Total etch resin based sealant ultraseal xt — Sealing deep pits and fissures
  Arms: Total-etch resin based sealant

SUMMARY:
The aim of the study is to clinically assess the effect of sandblasting prior to self-etch resin based sealant on its retention after one year follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have existing pits and fissures that are anatomically deep and caries susceptible.
* Stained pits and fissures with minimum decalcification of opacification and no softness at the base of the fissure (ICDAS 1 and 2).

Exclusion Criteria:

* An individual with no previous caries experience and well coalesced pits and fissures.
* Partially erupted teeth.

  * Teeth with cavitation or caries of the dentin.
* Teeth with dental fluorosis, Hypocalcification

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Retention rate | Change from baseline at 3, 6, 12 months
  •Full retention (FR): the material was fully present on the occlusal surfaces •Partially lost (PL): the material was present, but as a result of either wear or loss of the material, part of a previously sealed pit or fissure, or both, was exposed. •Totally lost (TL): no trace of the material was detected on the surface.

CONTACTS AND LOCATIONS:
Overall Officials: Rawda Hesham H. Abd ElAziz, Post Phd, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided